CLINICAL TRIAL: NCT05485532
Title: Development and Validation of a Telemonitoring System for High-risk Cardiovascular Patients
Acronym: TELE-CARDIO
Status: Active, not recruiting | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Univ. Prof. Dr. Axel Bauer, Director of Department for Internal Medicine III - Cardiology and Angiology, Medical University Innsbruck
Other Study IDs: 1282/2020
Record Dates: First submitted 2022-07-21; First posted 2022-08-03 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Telemonitoring System using Cosinuss° Two and/or Garmin Vivoactive 4 — Development and validation of a telemonitoring system using smart devices

SUMMARY:
Development and validation of a telemonitoring system for high-risk cardiovascular patients.

The main purpose of this study is to investigate the beneficial effect of continuous telemonitoring in patients with cardiovascular diseases in different clinical settings (hospitalized patients, ambulant patients, patients during cardiac rehabilitation,...) Beside established risk parameters such as HRV (heart rate variability) and DC (Deceleration Capacity) new risk stratification models should be established from the continuously recorded biosignals.

ELIGIBILITY:
Inclusion Criteria:

* decidable male and female patients > 18 years of age
* cardiovascular disease with at least one of the following criteria:
* LVEF ≤ 40%
* cardiac autonomic dysfunction
* St. p. myocardial infarction
* St. p. cardiopulmonary resuscitation
* St. p. pulmonalartery embolism
* St. p. decompensated heart failure
* Informed consent for participation in the clinical trial

Exclusion Criteria:

* missing informed consent
* pregnant and breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with presence of inclusion criteria presenting at one of the participating centres.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
occurence of combination of cardiovascular mortality, stroke, myocardial infarction and hospitalization due to decompensated heart failure | from inclusion to end of study (max. 3 years)

SECONDARY OUTCOMES:
occurence of all cause mortality | from inclusion to end of study (max. 3 years)
occurence of cardiovascular mortality | from inclusion to end of study (max. 3 years)
occurence of stroke | from inclusion to end of study (max. 3 years)
occurence of myocardial infarction | from inclusion to end of study (max. 3 years)
number of patients with hospitalization due to decompensated heart failure | from inclusion to end of study (max. 3 years)
number of patients with hospitalization due to other cardiovascular condition | from inclusion to end of study (max. 3 years)
number of patients admitted to intensive care unit | from inclusion to end of study (max. 3 years)
number of days with successful telemonitoring | from inclusion to end of study (max. 3 years)

OTHER OUTCOMES:
Cardiac Autonomic Function | from inclusion to end of study (max. 3 years)
  Heart Rate Variability (HRV), Deceleration Capacity (DC), Periodic Repolarization Dynamics (PRD), Baroreflex Sensitivity, ...

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - Medizinische Universität Innsbruck, Univ.-Klinik für Innere Medizin III, Kardiologie und Angiologie, Innsbruck, Tyrol
  - Reha Zentrum Münster, Münster, Tyrol

IPD SHARING:
Plan to Share IPD: No